CLINICAL TRIAL: NCT05385003
Title: An Interventional Study for the Beneficial Effects of Prebiotics on Hyperuricemia in Chinese Subjects
Brief Title: Effect of Prebiotics on Hyperuricemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pre-2022
Record Dates: First submitted 2022-05-13; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Subjects With Hyperuricemia
MeSH Terms: interventions — Anserine; SFTI-1 peptide, sunflower

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Supplement: anserine (Experimental): Subjects are instructed to take one capsule of anserine daily for a total of 3 months
  Interventions: Dietary Supplement: anserine
- Dietary Supplement: Sunflower peptide (Experimental): Subjects are instructed to take one capsule of Sunflower peptide daily for a total of 3 months
  Interventions: Dietary Supplement: Sunflower peptide
- Dietary Supplement: Placebo control (Placebo Comparator): Subjects are instructed to take one capsule of placebo daily for a total of 3 months
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: anserine — During the study period, subjects are instructed to take one capsule of anserine daily for a total of 3 months. Aside from the prebiotic supplement, all participants are instructed to continue their normal routine and not make any changes to their exercise habits but reduce purine intake.
  Arms: Dietary Supplement: anserine
Dietary Supplement: Sunflower peptide — During the study period, subjects are instructed to take one capsule of Sunflower peptide daily for a total of 3 months. Aside from the prebiotic supplement, all participants are instructed to continue their normal routine and not make any changes to their exercise habits but reduce purine intake.
  Arms: Dietary Supplement: Sunflower peptide
Dietary Supplement: Placebo control — During the study period, subjects are instructed to take one capsule of placebo control daily for a total of 3 months. Aside from the probiotic supplement, all participants are instructed to continue their normal routine and not make any changes to their exercise habits but reduce purine intake.
  Arms: Dietary Supplement: Placebo control

SUMMARY:
Hyperuricemia is a major risk factor for many chronic diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of Hyperuricemia. Animal studies have demonstrated that administration of prebiotics help delay the progression of Hyperuricemia through several mechanisms. This trial aims to examine its protective effect in humans.

DETAILED DESCRIPTION:
Hyperuricemia is a major risk factor for many chronic diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of hyperuricemia. Animal studies have demonstrated that administration of prebiotics help delay the progression of hyperuricemia through several mechanisms such as reduction in endotoxemia, and enhanced production of short-chain fatty acids.

However, whether administration of prebiotics also has a protective effect in subjects with Hyperuricemia remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* Local residents aged between 18-65 years old;
* Stable weight (<5% weight change over last 3 months);
* Fasting uric acid was > 420μmol/L for male and > 360μmol/L for female on two different days
* Those who have never taken uric acid lowering drugs or have stopped taking uric acid lowering drugs for at least four weeks;
* Absence of any diet or medication that might interfere with Uric acid metabolism and gut microbiota, especially antibiotics and probiotics at least 4 weeks before recruitment.

Exclusion Criteria:

* Acute illness or evidence of any acute or chronic inflammatory of infective diseases;
* Participation in regular diet program more than 2 times per week in the latest 3 months prior to recruitment;
* Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study.
* Women of childbearing age who are pregnant, breast-feeding or preparing for pregnancy; Patients who had surgery within the past six months or planned surgery during the trial period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum Uric acid | from baseline to 12 weeks after intervention
  change of fasting uric acid level assessed by biochemical detector
Change of excretion of uric acid | from baseline to 12 weeks after intervention
  excretion rate of uric acid assessed by secretion rate of uric acid in urine during 3 hours

SECONDARY OUTCOMES:
Change of Gut microbiota | from baseline to 12 weeks after intervention
  Alterations of the composition of gut microbiota evaluated by metagenomics
Change of Microbial metabolites | from baseline to 12 weeks after intervention
  Untargeted metabolomics will be used to assess the alterations of microbial metabolites with High performance liquid chromatography-mass spectrometry
Change in blood pressure | from baseline to 12 weeks after intervention
  Change in blood pressure assessed by electronic sphygmomanometer
Change in fasting glucose | from baseline to 12 weeks after intervention
  Change in fasting glucose assessed by biochemical detector
Change in waist circumference | from baseline to 12 weeks after intervention
  Change in waist circumference assessed by tape
Change in lipid profiles | from baseline to 12 weeks after intervention
  Change in total cholesterol, triglycerides, LDL-c and HDL-c assessed by biochemical detector

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Department of Nutrition and Food Hygiene, Guangzhou, Guangdong
  - Sun Yat-Sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No